CLINICAL TRIAL: NCT06079645
Title: Triamcinolone Acetonide Injections Compared With Micro Injections (MMP Technique) of Triamcinolone Acetonide for the Treatment of Female Genital Lichen Sclerosus and Atrophic
Brief Title: Lichen Sclerosus - Treatment With Triamcinolone Acetonide: Injections (Syringe and Needle) x Micro Injections (MMP Technique)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Dermatologica Arbache ltda (Other)
Responsible Party: Principal Investigator, SAMIR ARBACHE, PHD, Clinica Dermatologica Arbache ltda
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lichen Sclerosus of External Female Genital Organs
Keywords: acetonide, triamcinolone; Vulvar Diseases; Administration, Cutaneous; Syringes; Tattooing
MeSH Terms: conditions — Vulvar Diseases | interventions — Needles

STUDY DESIGN:
Intervention Model Description: Prospective, randomized pilot study involving 20 participants with genital LEA, refractory to the use of high-potency topical corticosteroid therapy. In this investigation.
  The vulvas will be randomized as right side and left side
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triamcinolone acetonide (2mg/ml) injections through syringes and needles (Active Comparator): Triamcinolone at a concentration of 2mg/ml will be injected on one side of the randomized vulva using a syringe and needle.
  Interventions: Procedure: Infiltration of triamcinolone acetonide (2mg/ml) through syringes and needles
- Triamcinolone acetonide (40mg/ml) through microinjections with needles (Active Comparator): Triamcinolone at a concentration of 40mg/ml will be injected on the other side of the randomized vulva using a tattoo machine.

INTERVENTIONS:
Procedure: Infiltration of triamcinolone acetonide (2mg/ml) through syringes and needles — Infiltration of triamcinolone acetonide (2mg/ml) through syringes and needles
  Arms: Triamcinolone acetonide (2mg/ml) injections through syringes and needles
Procedure: Infiltration of triamcinolone acetonide (40 mg/ml) with needles — Infiltration of triamcinolone acetonide (40 mg/ml) through needles of tattoo machine

SUMMARY:
This research is about a genital disease known as Lichem Sclerosus and Atrophic. It mainly affects women over 18 years of age. The treatment will involve injections of a medicine that contains cortisone, using two different methods: with a syringe and a needle or with a tattoo machine. Before and after treatment, they will see if women feel pain, itching, burning, scratching or difficulty having sexual intercourse.

DETAILED DESCRIPTION:
There is evidence that injectable triamcinolone has an effect on reducing the symptoms of lichen sclerosus and atrophic. After randomizing the vulva, the vulva will be anesthetized with lidocaine infiltrations. After 15 minutes, interventions will begin. Triamcinolone will be injected using two different techniques: syringes & needles in one side and with tattoo machine (MMP technique) in other side. The outcomes will be evaluated according to the criteria of pain, itching, burning, itching and difficulty in sexual penetration

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and/or histopathological diagnosis of genital (vulvar, perineal or perianal) Lichen Sclerosus and Atrophicus (LEA),
2. Failure to regress symptoms after topical treatment with potent topical corticosteroid for at least 3 months,
3. Progressive deformity of the vulva, clitoris, perineal or perianal region during treatment with potent topical corticosteroids,

Exclusion Criteria:

* Absence of other skin diseases such as lichen planus, psoriasis, Crohn's disease and ulcerative colitis,
* Commitment to use at least one form of adequate contraception (hormonal or barrier method) if sexually active or of childbearing potential (premenopausal or postmenopausal women for less than 2 years),
* Willingness to fulfill the study requirements. Willing and able to follow the schedule of treatments and follow-up visits,
* patient demonstrates mental and psychiatric health,
* Signs of good hygiene and evidence that you can apply dressings until the injuries heal,
* Diagnosis of pre-malignant or malignant genital (e.g. vulvar dysplasia, intraepithelial neoplasia or carcinoma),
* Crural lymphadenopathy,
* Absence of urinary incontinence, absence of immunological changes, absence of visceral neoplasia, absence of coagulation disorders (or use of anticoagulants), absence of immunosuppressive treatment (including) systemic corticosteroid therapy.
* Patients/participants with previously known allergies or those detected during the interventions (anesthetics, topical antibiotics or other medications used in the trials),
* If pregnancy occurs during the trial, the participant will be excluded from the investigation and referred to an obstetrician. If the patient wishes, her genitalia will be clinically monitored during pregnancy and breastfeeding,
* Participants who are not collaborative or who are absent from regular visits.
* Refusal to treat local infectious diseases that trigger intervention (parasitic, protozoal, bacterial, viral or fungal).
* Participant with recurrent genital herpes simplex who refuses to undergo systemic antiviral therapy.
* Identification during interventions of allergies to the medications used in the trial (anesthetics, topical antibiotics or other medications used in the trials),
* Any disease or condition not explicitly related to the exclusion criteria, which in the investigator's judgment interferes with the participant's ability to comply with the protocol, compromises the participant's safety or interferes with the interpretation of study results,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — treatment will only be carried out in women
Enrollment: 20 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-06-14 (Actual)

PRIMARY OUTCOMES:
Scoring System for Vulvar Lichen Sclerosus | one year
  On each side of the randomized vulva, symptoms of itching, burning, pain and dyspareunia will be assessed before and after the intervention. The assessment will be carried out by the patient herself, on a scale of zero to 10, with zero being asymptomatic and 10 when the symptom is unbearable.

SECONDARY OUTCOMES:
evaluate the safety of both interventions | one year
  ulcers, telangiectasias and local atrophies. Local or systemic infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Dermatologica Arbache Ltda, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be continuously shared with the Ethics Committee
Supporting Information: Study Protocol, CSR
Time Frame: 18 months
Access Criteria: reports will be sent continuously to the ethics committee

REFERENCES:
- [Background] Stucker M, Grape J, Bechara FG, Hoffmann K, Altmeyer P. The outcome after cryosurgery and intralesional steroid injection in vulvar lichen sclerosus corresponds to preoperative histopathological findings. Dermatology. 2005;210(3):218-22. doi: 10.1159/000083513. PMID 15785050
- [Background] Ventolini G, Swenson KM, Galloway ML. Lichen sclerosus: a 5-year follow-up after topical, subdermal, or combined therapy. J Low Genit Tract Dis. 2012 Jul;16(3):271-4. doi: 10.1097/LGT.0b013e31823da7e8. PMID 22258061
- [Background] Gunthert AR, Duclos K, Jahns BG, Krause E, Amann E, Limacher A, Mueller MD, Juni P. Clinical scoring system for vulvar lichen sclerosus. J Sex Med. 2012 Sep;9(9):2342-50. doi: 10.1111/j.1743-6109.2012.02814.x. Epub 2012 Jul 3. PMID 22759453
- [Background] Arbache S, Hirata SH. Efficacy and Safety of 5-Fluorouracil Tattooing to Repigment Idiopathic Guttate Hypomelanosis: A Split-Body Randomized Trial. Dermatol Surg. 2023 Jun 1;49(6):603-608. doi: 10.1097/DSS.0000000000003793. Epub 2023 Apr 3. PMID 37011024
- [Result] Mazdisnian F, Degregorio F, Mazdisnian F, Palmieri A. Intralesional injection of triamcinolone in the treatment of lichen sclerosus. J Reprod Med. 1999 Apr;44(4):332-4. PMID 10319301